CLINICAL TRIAL: NCT07052006
Title: A Phase 2a Study of HT-6184 in Subjects With IPSS-R Very Low, Low or Intermediate Risk Myelodysplastic Syndrome (MDS) and Symptomatic Anemia
Brief Title: A Phase 2a Study of HT-6184 in Subjects With IPSS-R Very Low, Low or Intermediate Risk MDS and Anemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Halia Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HT-6184-MDS-001; CTRI/2023/11/059758 (Other: Clinical Trials Registry - India)
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndrome; Anemia in Myelodysplastic Syndromes
Keywords: Very Low-risk MDS; Low-risk MDS; Intermediate-risk MDS; Symptomatic anemia
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HT-6184 (Experimental)
  Interventions: Drug: HT-6184

INTERVENTIONS:
Drug: HT-6184 — Oral HT-6184
  Other Names: Ofirnoflast

SUMMARY:
This research is being conducted to asses if HT-6184 is effective in the treatment of Very Low, Low, or Intermediate Risk Myelodysplastic Syndrome (MDS) and Symptomatic Anemia.

The study includes a 28-day Screening Period followed by a 16- or 32-week Treatment Period.

Participants will be monitored at each cycle for drug tolerance, safety, and hematological response. A response assessment will occur after 16 weeks of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Signed Informed Consent Form (ICF).
3. Adequate organ function.
4. A documented diagnosis of MDS or non-proliferative Myelodysplastic/myeloproliferative neoplasm (MDS/MPN).
5. Less than 10% bone marrow myeloblasts.
6. Refractory or intolerant of, or ineligible for treatment with an erythroid stimulating agent (ESA).
7. Prior ESA treatment must have been discontinued ≥ 2 weeks prior to date of study treatment.
8. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2.
9. Subjects must have symptomatic anemia.
10. Subjects with NGS (Next-generation sequencing) myeloid-specific somatic gene mutation profile with ≥ 5 % quantitation of clone size by variant allele frequency (VAF).
11. Women of child-bearing potential using an acceptable double-barrier method of contraception.
12. Male subjects who are using an acceptable method of contraception.

Exclusion Criteria:

1. Other causes of anemia such as iron deficiency.
2. Clinically significant anemia resulting from B12 or folate deficiencies, autoimmune or hereditary hemolysis, or gastrointestinal bleeding.
3. Women must not be pregnant or breastfeeding.
4. Presence of concomitant intercurrent illness which, in the opinion of the Investigator, would compromise safe participation in the study.
5. Secondary MDS.
6. Treatment with cytotoxic chemotherapeutic agents or experimental agents for the treatment of MDS within 4 weeks of study treatment.
7. Chronic use of systemic corticosteroids for comorbid or study disease condition within last 4 weeks of study treatment.
8. Prior history of malignancy other than MDS.
9. Subject has undergone a stem cell, bone marrow or solid organ transplant
10. Subjects with positive serology for Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or Human Immunodeficiency Virus (HIV).
11. Prior treatment with disease modifying agents.
12. Participation in any clinical study within 90 days before the first dose of Investigational Product.
13. Loss of ≥ 350 ml of blood within 90 days before the first dose of Investigational Product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-12-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The rate of hematological improvement. | 16 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- India (10):
  - Hemato Oncology Clinica Ahmedabad Pvt. Ltd. Vedanta Institute of Medical Sciences, Ahmedabad, Gujarat
  - Shalby Hospital, Ahmedabad, Gujarat
  - Malabar Cancer Center, Kannur, Kerala
  - HCG Cancer Center Vizag, Visakhapatnam, Krishna
  - Dr. Bafna's Star Superspeciality Clinic and Hospital, Kolhāpur, Maharashtra
  - All India Institute of Medical Sciences, Dehradun, Rishkesh
  - Meenakshi Mission Hospital and Research Centre, Madurai, Tamil Nadu
  - Apollo Cancer Centre, Hyderabad, Telangana
  - Nil Ratan Sircar Medical College and Hospital, Kolkata, West Bengal
  - Tata Medical Center, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No